CLINICAL TRIAL: NCT01010399
Title: A Pilot, Open-Label Study of Adjunctive Therapy With Lovaza® in Hypertriglyceridemic, HIV-Infected Subjects Who Switched Protease Inhibitor to Once-Daily Lexiva® 1400mg Plus Norvir® 100mg Plus Optimized Background
Brief Title: Boosted Lexiva With Lovaza Adjunctive Therapy in Hypertriglyceridemic, HIV-Infected Subjects
Acronym: BuLLET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Felizarta, Franco, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL112948
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-03

CONDITIONS: Hypertriglyceridemia; HIV Infection
Keywords: HIV; triglycerides; fosamprenavir
MeSH Terms: conditions — Hypertriglyceridemia; HIV Infections | interventions — Omacor; fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boosted Lexiva with Lovaza (Experimental)
  Interventions: Dietary Supplement: Lovaza; Drug: fosamprenavir/ritonavir

INTERVENTIONS:
Dietary Supplement: Lovaza — Lovaza at a dose of 4g per day with each 1g capsule containing 465 mg of eicosapentaenoic acid (EPA) and 375 mg of docosahexaenoic acid (DHA) for 18 weeks
Drug: fosamprenavir/ritonavir — Lexiva (fosamprenavir calcium) 1400 mg per day, Norvir (ritonavir) 100 mg per day

SUMMARY:
In subjects on boosted protease inhibitor (PI)-regimens who have elevated triglycerides, a switch to fosamprenavir/ritonavir once daily followed by the addition of Lovaza will result in 30% of patients achieving a reduction in fasting triglycerides < 200 mg /dL while maintaining virologic suppression.

ELIGIBILITY:
Inclusion Criteria:

* fasting triglycerides >= 200 mg/dL but <1,200 mg/dL
* fasting LDL <= 160 mg/dL
* participation in a lipid-lowering diet and exercise program for at least 28 days
* treatment with stable HAART consisting of first or second RTV-boosted PI regimen plus optimized background ART for at least 3 months
* plasma HIV-1 RNA <50 copies/mL
* CD4+ cell count >50 cells/mm3
* male subjection testosterone replacement therapy with total testosterone level <= 1 x upper limit of normal
* female study volunteer must use a form of contraception
* ability and willing ness to give written informed consent

Exclusion Criteria:

* any Grade 4 laboratory abnormality
* currently taking amprenavir or fosamprenavir
* required a second RTV-boosted PI for reasons of virologic failure
* atherosclerotic disease risk
* congestive heart failure (NYHA Class III or IV)
* uncontrolled hypertension
* history of pancreatitis
* active bleeding disorder
* recent history of significant renal, pulmonary, biliary, hepatic or gastrointestinal disease
* current diabetes mellitus requiring pharmacological treatment
* use of systemic cancer chemotherapy; active cancer
* pregnancy or breast-feeding
* requirement for any lipid-lowering agent after baseline
* use of hormonal anabolic therapies, systemic steroids, immune modulators
* use of anticoagulants, investigational antiretroviral drugs
* allergy to study drugs
* active CDC clinical category C event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Felizarta, MD, Principal Investigator — Franco Felizarta, MD
Locations (1):
- Franco Felizarta, MD, Bakersfield, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Boosted Lexiva With Lovaza
Started | 36
Completed | 31
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Boosted Lexiva With Lovaza
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Triglycerides <200 mg/dL
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Boosted Lexiva With Lovaza
Number analyzed (Participants) | 36
participants | 12

2. Secondary Outcome: Proportion of Subjects With HIV-1 RNA <50 Copies/mL
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Boosted Lexiva With Lovaza
Number analyzed (Participants) | 36
participants | 28

ADVERSE EVENTS:
Arm/Group | Boosted Lexiva With Lovaza
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 6/36
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boosted Lexiva With Lovaza (N=36)
hypercholesterolemia (Metabolism and nutrition disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 1 (1)
influenza (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes